CLINICAL TRIAL: NCT05616910
Title: Inhaled Nitric Oxide for Microvascular Dysfunction in Traumatic Brain Injury
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 851809
Record Dates: First submitted 2022-10-31; First posted 2022-11-15 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury
Keywords: hypoperfusion; cerebral blood flow; nitric oxide; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group iNO (Experimental): Subjects will receive iNO for 4 hours, followed by standard respiratory support (SRS) for 4 hours. This pattern will be reversed the next day (SRS then iNO). on the following day, the pattern will be reversed back to iNO for 4 hours and SRS for 4 hrs.
  Interventions: Drug: inhaled nitric oxide
- Group SRS (Sham Comparator): Subjects will receive standard respiratory support (SRS) for 8 hours.
  Interventions: Drug: inhaled nitric oxide

INTERVENTIONS:
Drug: inhaled nitric oxide — iNO will be provided by ventilator or nasal cannula for 4 hours each day.
  Other Names: standard respiratory therapy vs iNO

SUMMARY:
Traumatic brain injury (TBI) causes acute deficits in cerebral perfusion which may lead to secondary injury and worse outcomes. Inhaled nitric oxide (iNO) is a vasodilator that increases cerebral blood flow and is clinically used for hypoxic respiratory failure in neonates and adults. The investigators will perform a randomized controlled trial of iNO treatment in TBI patients acutely after injury. The investigators will then assess perfusion changes with optic neuromonitoring, blood biomarkers, and 6 month clinical outcomes.

DETAILED DESCRIPTION:
The objective of this study is to show that inhaled nitric oxide can increase blood flow in the brain after traumatic brain injury, attenuating brain injury and resulting in improved long-term function.

The investigators will use optical brain monitoring to determine changes in cerebral perfusion and metabolism by iNO treatment in TBI subjects. Within 24 hours of enrollment, TBI subjects meeting the inclusion criteria without exclusion criteria will undergo 8 hour sessions of monitoring (4 hours on iNO, 4 hours on standard respiratory therapy) for 4 days. During this time, Noninvasive Neuro-optic Monitoring (NNOM) device will be placed on the scalp and cerebral perfusion and metabolism parameters will be monitored to assess for therapeutic effect of iNO. There will be within-subject comparison of cerebral perfusion and metabolism on and off iNO. Also, there will be within-group comparison of cerebral perfusion and metabolism on days when iNO is given first vs days when iNO is given at a second session. Additionally, these parameters from this group will compared to a parallel group of TBI patients receiving 8 hours of only standard respiratory therapy for 4 days.

The investigators will assess the safety profile of iNO use in TBI subjects. During the course of iNO therapy in the initial 4 days, study subjects will be monitored for methemoglobinemia, hypotension, renal failure, neurological exam changes, and any other adverse events. Additionally, the investigators will assess blood-based biomarkers of injury with blood draws at the end of each iNO treatment session in TBI subjects for 4 days. During the initial 4 days of the trial, blood draws will be performed at the end of each session to detect biomarkers. Specifically, biomarkers that have been shown to correlate with injury severity such as GFAP, NFL, UCHL-1, tau, and S100B will be monitored at the end of iNO session and standard respiratory therapy session. This will be performed by using a novel assay termed SIMOA, a sensitive detection method for blood-based biomarkers.

As an exploratory aim, the investigators will compare 6-month GOS-E outcomes and injury biomarkers of the patients who received iNO to those who received standard respiratory therapy. Patients will be assessed for their functional status at the time of 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 (inclusive)
2. GCS 9-12 or GCS 13-15 with an abnormal imaging scan
3. Radiologic findings indicative of primarily diffuse TBI

Exclusion Criteria:

1. Severe cardiac dysfunction (e.g. elevation of pulmonary edema on chest xray, large elevation of cardiac enzymes)
2. Large focal injury (subdural hematoma, epidural hematoma, intraparenchymal hematoma, >30mL aggregate volume).
3. Need for immediate neurosurgical intervention
4. Pre-existing disabling psychiatric or neurological disorders such as cortical stroke, brain tumor, disabling multiple sclerosis, dementia, and severe TBI
5. Known intracranial vessel disease
6. Acute Respiratory Distress Syndrome (ARDS) or pre-existing pulmonary hypertension
7. Cardiopulmonary resuscitation or cardioversion at admission
8. Chronic Kidney Disease (Glomerular Filtration Rate <60mL/min/1.73m2)
9. Respiratory Infection
10. Prisoners, patients in police custody, pregnant women
11. Possible drug interactions (nitric oxide donors: prilocaine, sodium nitroprusside, nitroglycerin)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2028-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Cerebral Metabolism assessed by Spectroscopy | 4 days
  Metabolic Rate of oxygen consumption by the brain measured by diffuse correlation spectroscopy and time-resolved infrared-spectroscopy.

SECONDARY OUTCOMES:
Incidence of Inhaled Nitric Oxide induced methemoglobinemia | 4 days
  Methemoglobin levels of blood greater than 1%
Incidence of Inhaled Nitric Oxide induced hypotension | 4 days
  Blood pressure less than 90/60 mmHg for 30 minutes or longer
Incidence of Inhaled Nitric Oxide induced neurological deterioration | 4 days
  Glasgow coma scale decrease of 2 or more points.
Blood-based biomarkers of injury | 4 days, 6 months
  Levels of neurofilament-light, glial fibrillary acidic protein, tau, ubiquitin carboxy-terminal hydrolase L1 (all biomarkers are in units of pg/mL)
Long term functional outcome | 6 months
  Glasgow Outcome Scale Extended (GOS-E) (range: 1-8, 1: death, 8: good recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Shin, Principal Investigator — Assistant Professor
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No